CLINICAL TRIAL: NCT01997723
Title: Comparative Effectiveness Research to Enhance Outcomes in African-Americans With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bharati Prasad, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-0222; KM1CA156717 (NIH)
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA, portable monitoring, home diagnosis
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OSA testing (Experimental): Cross-over design, single group/arm Interventions: polysomnography with simultaneous portable monitoring and home portable monitoring administered to each participant in random order.
  Interventions: Device: Portable monitoring; Other: Polysomnography; Device: Home portable monitoring; Device: Laboratory portable monitoring

INTERVENTIONS:
Device: Portable monitoring — A device applied over 1 arm (on the wrist and finger), worn overnight by patients to detect OSA.
  Other Names: WatchPAT200, Itamar medical Inc.
Other: Polysomnography — One attended diagnostic sleep study.
Device: Home portable monitoring — Portable monitoring with WP200 device - applied by participants once at home.
Device: Laboratory portable monitoring — Portable monitoring with WP200 device - applied by technologist once in the laboratory simultaneously with polysomnography.

SUMMARY:
Obstructive Sleep Apnea (OSA) is under-diagnosed and is associated with increased cardiovascular morbidity and mortality. Laboratory-based overnight polysomnography (PSG) is the gold standard in clinical practice to diagnose OSA but has availability, cost, and resource limitations. In the last decade, an alternative diagnostic strategy, Portable Monitoring (PM) has emerged with the goal of reducing expense and delays in clinical management. In contrast to PSG, PM maybe performed unattended in homes, utilize different neurophysiologic and cardiorespiratory parameters, and may synthesize these data differently. PM is feasible and is approved by Centers for Medicare and Medicaid Services (CMS) in the United States. However, the diagnostic utility of PM in minority and underserved populations is not defined.

African-Americans are more severely affected by hypertension and cardiovascular disease (CVD) than other ethnic groups and OSA is more common in this population. OSA is a treatable cause of hypertension. Despite this the impact of timely interventions for OSA on health outcomes and risk reduction specific to African Americans is unknown.

Purpose of this research: In view of the vulnerability of this population and the potential for improvement in healthcare access for OSA with home-based diagnosis, this study aims to establish the feasibility and identify the potential advantages and limitations of home-based diagnosis of OSA in a high-risk urban African-American population including veterans with frequently limited access to healthcare.

Hypothesis: The investigators hypothesize that home-based PM is not inferior to standard laboratory-based PSG in effectively diagnosing OSA in urban African Americans.

DETAILED DESCRIPTION:
Hypothesis: The investigators hypothesize that home-based PM is not inferior to standard laboratory-based PSG in effectively diagnosing OSA in urban African Americans.

The specific aims of this project are:

Primary Aims: Aim 1. To compare the validity of a comprehensive and current PM technology to standard in-laboratory full PSG

1a) to measure and compare diagnostic accuracy of home-based PM with laboratory-PSG

1. b) to measure and compare diagnostic accuracy of simultaneous laboratory-based PM with laboratory-PSG Aim 2. To test the reliability and examine the applicability of PM in the home-setting
2. a) to compare diagnostic accuracy of home-based PM with laboratory-based PM

2b) to examine factors associated with technical reliability (data failure rate) of home-based PM 2c) to compare patient satisfaction and preference of testing in home-setting to laboratory-setting

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female African-Americans (age ≥18 years)
2. Berlin Questionnaire
3. Ability to understand written and verbal English

Exclusion Criteria:

1. Past treatment of OSA (medical, dental, or surgical)
2. Other primary sleep disorder(s) by history
3. Active uncontrolled medical conditions/immobility
4. Current drug or significant alcohol use
5. No current residential address or contact phone number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bharati Prasad, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Sleep Science Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Garg N, Rolle AJ, Lee TA, Prasad B. Home-based diagnosis of obstructive sleep apnea in an urban population. J Clin Sleep Med. 2014 Aug 15;10(8):879-85. doi: 10.5664/jcsm.3960. PMID 25126034

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Cross-over design, single group/arm
  Portable monitoring for OSA diagnosis: A device applied over 1 arm (on the wrist and finger), worn overnight by patients to detect OSA.
Period: Overall Study
Arm/Group | Experimental
Started | 75
Completed | 75
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Consenting adult men and women of self-identified African American ethnicity meeting inclusion/exclusion criteria were included.
Groups:
- OSA Testing: Cross-over design, single group/arm
  Interventions:
  One polysomnography one laboratory Portable monitoring simultaneously with polysomnography one home Portable monitoring
Arm/Group | OSA Testing
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 75
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
employed [Number; unit: participants] — 36/75 were employed, 39/75 were umemployed.
  participants | 36
Household income less than $50,000 per year [Number; unit: participants] — 57/75 had household income < $50,000 per annum and 18 had household income >/= $50,000 per annum
  participants | 57
Education less than or equal to high school [Number; unit: participants] — 26/75 had </=high school education and 49/75 had one or more years of college education.
  participants | 26

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI)
Description: AHI is the number of abnormal respiratory events (apneas and hypopneas) per hour of sleep.
  AHI on home portable monitor (PM) compared to AHI on laboratory polysomnography (PSG).
Time Frame: 4 days
Population: The polysomnography area under the curve (AUC) in an ROC plot for this study was assumed to be 0.99. The AUC for home PM test was targeted at 0.88 based on published report for power of 0.90 in a population with estimated pretest probability of 75-85%, ascertained by Berlin Questionnaire.
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- OSA Testing: Cross-over design, single group/arm
  Portable monitoring for OSA diagnosis: A device applied over 1 arm (on the wrist and finger), worn overnight by patients to detect OSA.
Arm/Group | OSA Testing
Number analyzed (Participants) | 75
events per hour
  Polysomnography AHI | 30.3 (35)
  Home Portable monitor AHI | 32.3 (27.6)
  Lab portable monitor AHI | 39.1 (29.1)

2. Secondary Outcome: Technical Failure Rate
Description: home PM tests that failed to provide technically adequate data for diagnosis. Technical failure(s) were tests where estimated total sleep time (TST) was ≤ 2 hours or portable monitor data of interpretable quality was less than 4 hours per recording.
Time Frame: 4 days
Measure: Number; unit: percentage of recordings
Arm/Group | OSA Testing
Number analyzed (Participants) | 75
percentage of recordings
  Home PM | 5.3
  Lab PM | 3.1

3. Other Pre Specified Outcome: Percentage of Participants Who Prefer Home Testing Over Laboratory Testing
Description: The participants indicated if they preferred Home Testing or in-laboratory Testing.
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | OSA Testing
Number analyzed (Participants) | 75
percentage of participants | 82

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | OSA Testing
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

LIMITATIONS AND CAVEATS:
This trial did not compare different portable devices for diagnostic accuracy compared to polysomnography (gold standard).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No